CLINICAL TRIAL: NCT01458119
Title: An Open-Label Extension Study to Evaluate the Long-Term Safety and Efficacy of Migalastat Hydrochloride Monotherapy in Subjects With Fabry Disease
Brief Title: Open-Label Phase 3 Long-Term Safety Study of Migalastat
Acronym: AT1001-041
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Amicus Therapeutics discontinued Study AT1001-041 for logistical reasons.
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT1001-041; 2011-004800-40 (EudraCT Number)
Record Dates: First submitted 2011-10-20; First posted 2011-10-24 (Estimated); Results first posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Fabry Disease
Keywords: Amicus Therapeutics; AT1001; Galafold; Migalastat
MeSH Terms: conditions — Fabry Disease | interventions — migalastat; larazotide acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Migalastat (Experimental): Migalastat 150-mg capsule taken orally QOD. The median duration of exposure was 23.5 m.
  Interventions: Drug: migalastat hydrochloride

INTERVENTIONS:
Drug: migalastat hydrochloride — Oral capsule QOD
  Other Names: AT1001; Galafold; Migalastat

SUMMARY:
This was a long-term, open-label study of migalastat (123 milligrams [mg] of migalastat [equivalent to 150 mg of migalastat hydrochloride]) (migalastat) in participants with Fabry disease who completed treatment in a previous monotherapy trial with migalastat.

DETAILED DESCRIPTION:
Study AT1001-041 was an open-label, noncomparative, multicenter, long-term extension study for participants with Fabry disease who completed treatment in one of three previous trials of migalastat (AT1001-011 [NCT00925301], AT1001-012 [NCT01218659], or FAB-CL-205 [NCT00526071]). In these trials, migalastat was given as monotherapy. This was an extension study designed to evaluate the long-term safety and efficacy of migalastat for the treatment of Fabry disease. Study visits occurred every 6 months (m). Visit evaluations included physical examinations, clinical laboratory parameters, adverse events, and participant reported outcomes.

The study consisted of a Baseline Visit, which was performed at the time of the final visit of the previous study, followed by clinic visits every 6 m for each year of the study. Study assessments included a physical examination, echocardiography, laboratory parameters, and participant-reported outcomes. Since participants enrolled in the study at varying time points based on the completion of the preceding migalastat study, treatment duration varied among participants. No maximum treatment duration was defined. There were no control groups in this study; all participants received migalastat as a 150-mg capsule taken orally once every other day (QOD) and inactive reminder capsules on alternate days.

The sponsor (Amicus Therapeutics) discontinued Study AT1001-041 for logistical reasons and not due to either safety concerns or lack of efficacy. For participants who were ongoing in Study AT1001-041 at the time of discontinuation, the investigators were offered participation in a similar open-label, long-term migalastat treatment study (AT1001-042 [NCT02194985]) for participants ongoing at discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Completed migalastat treatment in a previous Fabry disease protocol
* Both male and female participants were enrolled
* Age 16 years or older
* Male and female participants had to agree to use protocol-identified acceptable contraception

Exclusion Criteria:

* Estimated glomerular filtration rate (eGFR) in the previous study was <30 milliliters/minute/1.73 square meters (mL/min/1.73 m^2) unless there was a measured GFR available within 3 m of the Baseline Visit that was >30 mL/min/1.73 m^2
* Had undergone, or was scheduled to undergo, kidney transplantation or was currently on dialysis
* Pregnant or breast feeding
* Treated with another investigational drug (except migalastat) within 30 days of study start
* Unable to comply with study requirements, or deemed otherwise unsuitable for study entry, in the opinion of the investigator
* Had documented transient ischemic attack, stroke, unstable angina, or myocardial infarction within the 12 m before the Baseline Visit
* Had clinically significant, unstable cardiac disease in the opinion of the investigator
* Had a history of allergy or sensitivity to migalastat (including excipients) or to other iminosugars
* Required treatment with Glyset (miglitol) or Zavesca (miglustat)
* Had any intercurrent illness or condition that may have precluded the participant from fulfilling the protocol requirements
* Had a severe or unsuitable concomitant medical condition
* Had a clinically significant abnormal laboratory value and a clinically significant electrocardiogram finding at the Baseline Visit.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2011-10-14 (Actual); Primary Completion 2016-02-17 (Actual); Study Completion 2016-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Clinical Research, Study Director — Amicus Therapeutics
Locations (25):
- United States (11):
  - Atlanta, Georgia
  - Chicago, Illinois
  - Kansas City, Kansas
  - Boston, Massachusetts
  - Grand Rapids, Michigan
  - New York, New York
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Dallas, Texas
  - Fairfax, Virginia
  - Seattle, Washington
- Pilar, Argentina
- Australia (2):
  - Adelaide
  - Parkville
- Edegem, Belgium
- Porto Alegre, Brazil
- Montreal, Canada
- Copenhagen, Denmark
- Cairo, Egypt
- Garches, France
- Roma, Italy
- Barcelona, Spain
- Ankara, Turkey (Türkiye)
- United Kingdom (2):
  - London
  - Salford

REFERENCES:
- [Derived] Germain DP, Hughes DA, Nicholls K, Bichet DG, Giugliani R, Wilcox WR, Feliciani C, Shankar SP, Ezgu F, Amartino H, Bratkovic D, Feldt-Rasmussen U, Nedd K, Sharaf El Din U, Lourenco CM, Banikazemi M, Charrow J, Dasouki M, Finegold D, Giraldo P, Goker-Alpan O, Longo N, Scott CR, Torra R, Tuffaha A, Jovanovic A, Waldek S, Packman S, Ludington E, Viereck C, Kirk J, Yu J, Benjamin ER, Johnson F, Lockhart DJ, Skuban N, Castelli J, Barth J, Barlow C, Schiffmann R. Treatment of Fabry's Disease with the Pharmacologic Chaperone Migalastat. N Engl J Med. 2016 Aug 11;375(6):545-55. doi: 10.1056/NEJMoa1510198. PMID 27509102

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighty-five eligible participants with Fabry disease who completed treatment with migalastat in one of three previous studies (AT1001-011 [NCT00925301], AT1001-012 [NCT01218659], or FAB-CL-205 [NCT00526071]) were enrolled in this open-label extension study to enable the collection of long-term safety and efficacy data.
Groups:
- Migalastat: Participants received migalastat hydrochloride (migalastat) 150-milligram (mg) capsule (equivalent to 123 mg of migalastat) given orally once every other day (QOD) for a median duration of 23.5 months (m). Participants received an inactive reminder capsule on alternate days during the study.
Period: Overall Study
Arm/Group | Migalastat
Started | 85
Received at Least 1 Dose of Study Drug | 85
Safety Population | 85
Intent to Treat (ITT) Population (Received at least 1 dose of study drug.) | 85
ITT-Amenable Population (Amenable mutations based on Good Laboratory Practice (GLP) Human Embryonic Kidney (HEK) assay.) | 68
Completed | 65
Not Completed | 20
Not completed — Physician Decision | 4
Not completed — Withdrawal Due to Nonamenable Mutation | 1
Not completed — Pregnancy | 1
Not completed — Death | 2
Not completed — Adverse Event | 1
Not completed — Consent Withdrawn by Participant | 8
Not completed — Non-compliance With Study Drug | 3

BASELINE CHARACTERISTICS:
Population: ITT Population: All participants who received at least 1 dose of study drug after they enrolled into this open-label extension study.
Groups:
- Migalastat: Participants received migalastat 150-mg capsule given orally QOD for a median duration of 23.5 m. Participants received an inactive reminder capsule on alternate days during the study.
Arm/Group | Migalastat
Number analyzed (Participants) | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (12.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 33

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants Experiencing Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered migalastat that did not necessarily have a causal relationship with the treatment. Each AE was recorded at the time of reporting; visits typically occurred every 6 months. A TEAE was defined as an AE starting on or after the first study drug administration date. Serious AEs were life-threatening or resulted in death, persistent or significant incapacitation, inpatient or prolonged hospitalization, or a congenital anomaly. The criteria for AE severity were: Mild: minimal discomfort, does not interfere with normal everyday activities; Moderate: sufficiently discomforting, interferes with normal everyday activities; Severe: prevents normal everyday activities. The number of participants experiencing TEAEs is presented for those who received migalastat treatment. A summary of serious and all other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline to End of Follow-up (30 days after the end of this 42-month study), with AE reporting occurring at each study visit, which occurred once every 6 months.
Population: Safety Population: All participants who received at least 1 dose of study drug after they enrolled into this open-label extension study.
Measure: Number; unit: participants
Arm/Group | Migalastat
Number analyzed (Participants) | 85
participants
  Participants with at least 1 TEAE | 74
  Participants with at least 1 serious TEAE | 22
  Participants discontinued due to TEAEs | 1
  Participants with adverse events leading to death | 2
  Participants with TEAEs related to study drug | 14
  Participants with TEAEs unrelated to study drug | 60
  Participants with at least 1 mild TEAE | 22
  Participants with at least 1 moderate TEAE | 40
  Participants with at least 1 severe TEAE | 12

2. Secondary Outcome: Annualized Rate Of Change In The Estimated Glomerular Filtration Rate (eGFR)
Description: The annualized rate of change of the eGFR was assessed per participant by the slope of the simple linear regression between the observed values and the assessment times. It was calculated by using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation (eGFR [CKD-EPI]) and the Modification of Diet in Renal Disease (MDRD) equation (eGFR [MDRD]). The equations are as follows:
  eGFR [MDRD] = 175 * (Serum Creatinine)^-1.154 * (Age)^-0.203 * 1.212 (if black or African American) * 0.742 (if female); eGFR [CKD-EPI] = 141 * min(serum creatinine/kappa,1)^alpha * max(serum creatinine/kappa, 1)^-1.209 * 0.993^age * 1.1018(if female) * 1.159(if black or African American), where kappa is 0.7 for females and 0.9 for males, alpha is -0.329 for females and -0.411 for males, min is minimum of serum creatinine/kappa or 1, and max is the maximum of serum creatinine/kappa or 1. The number of participants with at least a Baseline and a post-Baseline value are presented.
Time Frame: Baseline, Every 6 m until the End of Study (42 m)
Population: ITT-Amenable Population: All participants who received at least 1 dose of study drug. Participants with mutant forms of α-Galactosidase (Gal) A determined to be amenable to migalastat based on the GLP-HEK assay are referred to as "with amenable mutations." Number of participants analyzed are those with at least a Baseline and a post-Baseline value.
Measure: Mean (95% Confidence Interval); unit: milliliters/minute/1.73 meters^2
Groups:
- Migalastat ITT-Amenable Population: Participants received migalastat 150-mg capsule given orally QOD for a median duration of 23.5 m. Participants received an inactive reminder capsule on alternate days during the study. The ITT-amenable population included all participants who received at least 1 dose of study drug after they enrolled into this open-label extension study. Participants with mutant forms of α-Gal A determined to be amenable to migalastat treatment based on the GLP-HEK assay are referred to as "with amenable mutations."
Arm/Group | Migalastat ITT-Amenable Population
Number analyzed (Participants) | 47
milliliters/minute/1.73 meters^2
  EGFR [CKD-EPI] | 1.54 [-1.63 to 4.71]
  eGFR [MDRD] | 1.40 [-3.14 to 5.94]

ADVERSE EVENTS:
Time Frame: Baseline to End of Follow-up (30 days after the end of this 42-month study), with AE reporting occurring at each study visit, which occurred once every 6 months.
Arm/Group | Migalastat
Serious Adverse Events (participants affected / at risk) | 22/85
Other Adverse Events (participants affected / at risk) | 57/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Migalastat (N=85)
Implantable defibrillator insertion (Surgical and medical procedures) | 2
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Death (General disorders) | 1
Device malfunction (General disorders) | 1
Conversion disorder (Psychiatric disorders) | 1
Priapism (Reproductive system and breast disorders) | 1/33
Uterine polyp (Reproductive system and breast disorders) | 1/52
Foot fracture (Injury, poisoning and procedural complications) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Brain stem ischaemia (Nervous system disorders) | 1
Hemiplegic migraine (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Hepatic infarction (Hepatobiliary disorders) | 1
Calculus urinary (Renal and urinary disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Thyroid mass (Endocrine disorders) | 1
Pneumonia (Infections and infestations) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Migalastat (N=85)
Hypertension (Vascular disorders) | 6
Contusion (Injury, poisoning and procedural complications) | 5
Atrial fibrillation (Cardiac disorders) | 7
Palpitations (Cardiac disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Headache (Nervous system disorders) | 11
Dizziness (Nervous system disorders) | 9
Paraesthesia (Nervous system disorders) | 5
Fatigue (General disorders) | 9
Oedema peripheral (General disorders) | 6
Pain (General disorders) | 5
Pyrexia (General disorders) | 7
Vertigo (Ear and labyrinth disorders) | 5
Anxiety (Psychiatric disorders) | 5
Abdominal distension (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 11
Back pain (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11
Influenza (Infections and infestations) | 9
Nasopharyngitis (Infections and infestations) | 9
Upper respiratory tract infection (Infections and infestations) | 6
Urinary Tract Infection (Infections and infestations) | 8

LIMITATIONS AND CAVEATS:
The study was discontinued for logistical reasons and not due to either safety concerns or lack of efficacy. The investigators were offered participation in a similar long-term migalastat study for participants ongoing at discontinuation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator can publish only the results from this trial, provided they supply the sponsor (or authorized entity) a copy of any proposed publication for review prior to submission for publication. If requested and prior to publication, the investigator will remove information deemed confidential or proprietary by the sponsor and will withhold publication an additional period of time to allow the sponsor to take appropriate measures to establish and preserve its proprietary rights.